CLINICAL TRIAL: NCT02930187
Title: Agreement Between Disease Activity and Ultrasound Scoring (Naredo-12) in Patients With Rheumatoid Arthritis With Clinical Remission in Daily Practice.
Brief Title: Ultrasound Evaluation of Remission in Rheumatoid Arthritis
Acronym: EVER-1
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC14.258; DR-2015-072 (Other: CNIL)
Record Dates: First submitted 2016-09-09; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis Patient With Remission :Ultrasonographic Disease Activity
Keywords: Rheumatoid arthritis, remission, ultrasound
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate correlations between the validated 12 joints-Naredo ultrasound score (B-mode (0-3), PD (0-3) or PDUS (0-3, max between B-mode or PD)) and the DAS28-ESR, DAS28-CRP, CDAI, SDAI and ACR-EULAR criteria for remission in routine care.

DETAILED DESCRIPTION:
Clinical remission is now a realistic goal in managing rheumatoid arthritis (RA) with treat to target strategy assessed according to different composite scores (DAS28, Simplified Disease Activity Index (SDAI), Clinical Disease Activity Index (CDAI), ACR-EULAR 2011 for remission). There are, however, no validated ultrasound remission criteria because of continuing uncertainty on the signification of persistent synovial hypertrophy in B-mode or Power Doppler (PD) mode in RA patients in clinical remission.

The objective was to evaluate correlations between the validated 12 joints-Naredo ultrasound score (B-mode (0-3), PD (0-3) or PDUS (0-3, max between B-mode or PD)) and the DAS28-ESR, DAS28-CRP, CDAI, SDAI and ACR-EULAR criteria for remission in routine care.

This french multicenter cross-sectional study took place in 11 rheumatology departments. The inter and intra-observer reproducibility for the ultrasound scoring was good to excellent. Inclusion criteria were as follows: RA meeting ACR-EULAR criteria, <15 years of progression, DAS-28-ESR<2.6 for at least 3 months, with a stable treatment including corticoids if necessary (equivalent prednisone<0.1 mg/kg) for 6 months. A standardized US examination was performed by an experience ultrasonographist blinded to clinical data. Spearman's correlation coefficients were determined between the Naredo12 B-mode (min-max,0-36), PD mode (0-36) and PDUS (0-36) scores and the different clinical remission scores. The impact of disease duration or duration of the clinical remission on ultrasound scores was also assessed (Kruskall-Wallis's test).

ELIGIBILITY:
Inclusion Criteria:

* Adults (âged of 18 or more),
* Rheumatoid arthritis according to ACR-EULAR 2010 criteria, during less than 10 years at least
* Remission according to DAS28-VS (<2.6) since 3 months at least,
* Disease modifying anti-rheumatic drugs and/or biotherapy stable dose since 6 months at least
* Steroids ≤0.1 mg/kg/day without high dose during the last 3 months
* Oral and written information and consent

Exclusion Criteria:

* Patient participating to a clinical trial about rheumatoid arthritis treatment
* Patient under administrative supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis in Routine Care
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
correlation between ultrasonography score Naredo12 B-mode and disease activity score (DAS28, SDAI, CDAI) | august 2015-april 2016
  Composit outcome measure : Ultrasonography score PD mode (0-36) Disease activityscore DAS28-ESR (0-10) Disease activity score DAS28-CRP (0-10) Disease activity score SDAI (0-86) Disease activity score CDAI (0-76)

SECONDARY OUTCOMES:
Correlation between ultrasonographic score PD mode and disease activity scores (DAS28, SDAI, CDAI). | august 2015-april 2016
  Composit outcome measure : Ultrasonography score PD mode (0-36) Disease activityscore DAS28-ESR (0-10) Disease activity score DAS28-CRP (0-10) Disease activity score SDAI (0-86) Disease activity score CDAI (0-76)
Correlation between ultrasonography scores PDUS and disease activity scores (DAS28, SDAI, CDAI). | august 2015-april 2016
  Composit outcome measure : Ultrasonography score PD mode (0-36) Disease activityscore DAS28-ESR (0-10) Disease activity score DAS28-CRP (0-10) Disease activity score SDAI (0-86) Disease activity score CDAI (0-76)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gaudin, Pr, Principal Investigator — University Hospital, Grenoble

REFERENCES:
- [Background] Aletaha D, Ward MM, Machold KP, Nell VP, Stamm T, Smolen JS. Remission and active disease in rheumatoid arthritis: defining criteria for disease activity states. Arthritis Rheum. 2005 Sep;52(9):2625-36. doi: 10.1002/art.21235. PMID 16142705
- [Background] Aletaha D, Smolen JS. The Simplified Disease Activity Index (SDAI) and Clinical Disease Activity Index (CDAI) to monitor patients in standard clinical care. Best Pract Res Clin Rheumatol. 2007 Aug;21(4):663-75. doi: 10.1016/j.berh.2007.02.004. PMID 17678828
- [Background] Ozgocmen S, Ozdemir H, Kiris A, Bozgeyik Z, Ardicoglu O. Clinical evaluation and power Doppler sonography in rheumatoid arthritis: evidence for ongoing synovial inflammation in clinical remission. South Med J. 2008 Mar;101(3):240-5. doi: 10.1097/SMJ.0b013e318164e16a. PMID 18364651
- [Background] Balsa A, de Miguel E, Castillo C, Peiteado D, Martin-Mola E. Superiority of SDAI over DAS-28 in assessment of remission in rheumatoid arthritis patients using power Doppler ultrasonography as a gold standard. Rheumatology (Oxford). 2010 Apr;49(4):683-90. doi: 10.1093/rheumatology/kep442. Epub 2010 Jan 4. PMID 20047979
- [Background] Saleem B, Brown AK, Keen H, Nizam S, Freeston J, Wakefield R, Karim Z, Quinn M, Hensor E, Conaghan PG, Emery P. Should imaging be a component of rheumatoid arthritis remission criteria? A comparison between traditional and modified composite remission scores and imaging assessments. Ann Rheum Dis. 2011 May;70(5):792-8. doi: 10.1136/ard.2010.134445. Epub 2011 Jan 17. PMID 21242236